CLINICAL TRIAL: NCT04847817
Title: Important Data on COVID-19 Profile in Africa
Acronym: AIDCO
Status: Completed | Type: Observational
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Leiden University Medical Center (Other); Institut de recherche en santé de surveillance épidémiologique et de formation (Unknown); Université des Sciences de la Santé (Unknown); Armauer Hansen Research Institute, Ethiopia (Other); Universität Tübingen (Other)
Responsible Party: Sponsor
Other Study IDs: 0011/2020/PR/SG/CNE; CEI-10/2020 (Other: Comité d'Ethique Institutionnel)
Record Dates: First submitted 2020-10-16; First posted 2021-04-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus Infection; Africa
Keywords: Coronavirus infection; SARS-CoV; COVID-19; Transmission; Africa
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal mucosal Blood Urine Stool

GROUPS / COHORTS (2):
- Index cases: Patients infected by SARS-Cov2 Polymerase Chain Reaction (PCR) and hospitalized in a referral center for COVID-19 .
- Households cases: Household contacts of SARS-Cov2 hospitalized COVID-19 patients.

SUMMARY:
The purpose of this study is to Understand the natural history of Coronavirus 2019 (COVID-19) infection to better define the period of infectiousness and transmissibility and to establish biobanks of COVID-19 blood and mucosal samples.

DETAILED DESCRIPTION:
In this study ,the participants will be enrolled sequentially in the COVID-19 care referral centers. The infected hospitalized patient will be identified by the physicians in hospital. After the patient has given his/her informed consent the permission will be sought from him to approach his household contacts. The household contacts will be screened, and included in the study.

Patients hospitalized and positive for COVID-19 by PCR and their household contacts of all ages and gender (40% minimum of female), will be enrolled upon receipt of written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Molecular (PCR) confirmed COVID-19 patients hospitalized in referral centers,
* Household contacts of hospitalized COVID-19 patient,
* Provided signed informed consent.

Exclusion Criteria:

* Pregnancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of volunteer COVID-19 patients hospitalized in referral center for COVID-19 care as well as the household contacts of these hospitalized COVID-19 patients in Gabon, Senegal and Ethiopia.
Sampling Method: Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
clinical and biological parameters of COVID-19 | 14 days
  Infection and disease progression - Pattern of virus transmission
SARS-CoV-2 transmissibility | 14 days
  proportion of household contact who will become positive for SARS-COV2 using PCR

CONTACTS AND LOCATIONS:
Overall Officials: Ayôla Akim ADEGNIKA, Principal Investigator — Centre de Recherches Médicales de Lambaréné; Marielle BOUYOU-AKOTET, Principal Investigator — Université des Sciences de Santé
Locations (2):
- Gabon (2):
  - Centre de Recherches Médicales de Lammbaréné, Lambaréné, Moyen-Ogooué Province
  - Centre de Recherches Médicales de Lambréné, Lambaréne

IPD SHARING:
Plan to Share IPD: Yes
Results from our COVID-19 AFRICA, AIDCO, project will be published in peer reviewed journals, seeking rapid and open access publication. This will be done as fast and widely as possible. Results will also be submitted and presented in any national, regional and international scientific meetings and congresses dedicated to COVID-19 online or face to face if, permitted. Before submission for publication or presentation, the review process outlined in the Consortium Agreement and agreed upon by all partners will be followed and care will be taken with respect to intellectual property protection.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years